CLINICAL TRIAL: NCT00563511
Title: A Randomized Controlled Trial on Smoking Cessation and Adherence Intervention on Patients With Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The University of Hong Kong (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: EC1966-02; HARECCTR0500052; HKU7428/03M
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Smoking Cessation
Keywords: smoking cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Methods

INTERVENTIONS:
Procedure: adherence intervention
Procedure: intervention without adherence advice
Procedure: control

SUMMARY:
The purpose of this proposed RCT is to test (a) the effectiveness of smoking cessation intervention (counseling and NRT) among patients with ED; and (b) the effectiveness of adherence intervention (ADIN) to increase adherence to NRT use in order to increase quit rate.

ELIGIBILITY:
Inclusion Criteria:

* Male ethnic Chinese aged 18 or above
* Smokes at least 1 cigarette per day
* Is not following other forms of smoking cessation interventions
* Intends to quit smoking within the next 7 days of the first contact and would use NRT
* Free from illness that contraindicate to the use of NRT
* Has signed an informed consent form, or has given verbal consent (for those contacted by telephone)

Exclusion Criteria:

* Patients who are psychologically or physically unable to communicate
* Children and teenagers (aged below 18)
* Those on regular psychotropic medications and in the presence of any serious health problems that may make them unsuitable for using NRT, such as recent stroke, palpitation, or other life threatening conditions

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Enrollment: 1210 (Estimated)
Dates: Start 2004-01; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
quit rate | 6-month
adherence rate | 4-weeks after the first use of NRT

SECONDARY OUTCOMES:
erectile function | 6-month
use of NRT | 3-month
quit rate | 3-month

CONTACTS AND LOCATIONS:
Overall Officials: TH Lam, Prof, Principal Investigator — Department of Community Medicine, The University of Hong Kong
Locations (4):
- China (4):
  - HKFPA, Hong Kong
  - Kwong Wah Hospital, Hong Kong
  - The University of Hong Kong, Hong Kong
  - WHO, Hong Kong